CLINICAL TRIAL: NCT03324165
Title: Randomized Control Trial Comparing Proposed Algorithm and Current Best Practice in the Evaluation of Suspected Appendicitis
Brief Title: Comparing Proposed Algorithm and Current Practice in the Evaluation of Suspected Appendicitis
Acronym: RCTAppAlg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Sengkang Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CIRB 2015/2981; NMRC/HSRNIG/0012/2015 (Other Grant/Funding Number: National Medical Research Council (NMRC), Singapore)
Record Dates: First submitted 2017-10-05; First posted 2017-10-27 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Acute Appendicitis
Keywords: Computed Tomography; Algorithm; Alvarado Score
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Arm (No Intervention): Patients randomized to Usual Care Arm will be managed as per current best practice that is based on the individual doctor's discretion.
- Intervention Arm (Experimental): Patients randomized to Intervention Arm will be managed as per the proposed algorithm, which is based on the computation of Alvarado Score.
  Interventions: Other: Proposed Algorithm

INTERVENTIONS:
Other: Proposed Algorithm — Proposed algorithm that uses Alvarado Score to guide CT utilization
  Arms: Intervention Arm

SUMMARY:
Acute appendicitis is one of the most common causes of acute abdominal pain requiring surgical intervention. In the current era, with diagnostic imaging technique like Computed Tomography (CT), negative appendectomy rates have been greatly reduced. However, the radiation risk with CT poses as a concern. Rules for clinical decision guiding CT utilization is thus essential to minimize unnecessary CT scans, which not only poses a radiation risk but also contributes to increased healthcare costs.

Through the development of an algorithm based on Alvarado Score for the management of acute appendicitis, investigators hope to reduce CT utilization with an acceptable negative appendectomy rate, and hence reducing unnecessary radiation and the healthcare costs involved.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common causes of acute abdominal pain requiring surgical intervention, with a lifetime risk of 8.6% for males and 6.7% for females. Historically, negative appendectomy rates of more than 20% were considered the norm. This is no longer acceptable in the current era, as despite low complication rates in the setting of negative appendectomy, conditions such as incisional hernias, intestinal obstruction secondary to adhesions and stump leakages can still result in significant morbidity.

Computed Tomography (CT) scan has emerged as the dominant imaging modality for evaluation of suspected appendicitis in adults. It has decreased negative appendectomy rates to fewer than 10%. However, the radiation exposure with CT poses a concern, particularly in appendicitis, which occurs predominantly in young patients most susceptible to the adverse effects of radiation. Available literature has estimated that at least 25% of CT scans are not clinically warranted and may pose more harm than benefits. Rules for clinical decision guiding CT utilization is thus essential to minimize unnecessary CT scans, which not only poses a radiation risk but also contributes to increased healthcare costs.

Currently, the management of suspected appendicitis is surgeon dependent. Accuracy of diagnosis is dependent on individual's clinical acumen, preference for CT scan and threshold for offering surgery. There is also a recent trend towards indiscriminate CT utilization with an estimated 1 in 4 CT scans ordered found to be clinically unwarranted. The Alvarado Score (AS) is a 10 point clinical scoring system for acute appendicitis that has been extensively validated. AS on a prospective database of 500 consecutive cases of suspected appendicitis admitted to Singapore General Hospital, Department of General Surgery from August 2013 to July 2014, was validated. A comparison was then made between diagnostic performance measures of CT scan and AS to identify ranges of AS where patients are unlikely to benefit from CT evaluation. From these findings, an objective algorithm for the management of suspected appendicitis guided by AS was formulated. Ideally, the algorithm will streamline CT utilization and reduce the number of CT scans ordered with an acceptable negative appendectomy rate. Thus, investigators hope to validate this proposed algorithm through a randomized control trial.

The trial will recruit 160 eligible patients over 2 years. Eligible patients who consented to participate in the trial will be subjected to randomization into one of the two trial groups - Usual Care Arm or Intervention Arm - in equal numbers (n=80). Patients randomized to Usual Care Arm will be managed according to individual's doctor discretion. On the other hand, patients randomized to Intervention Arm will have their Alvarado Score tabulated and managed as per proposed algorithm.

The primary objective of the trial is to show that the proposed management algorithm is effective in reducing the percentage of CT utilization as compared to current best practice for patients with suspected appendicitis seen at Singapore General Hospital and Sengkang Health. The hypothesis is that the proposed management algorithm will reduce the percentage of CT scans from 80%, which is the CT utilization rate when current best practice is used, to 60%. The study will be powered to detect this decrease with a 5% type I error rate.

The secondary objective of the trial is to estimate the proportion of negative appendectomy and missed diagnosis in each of the study arm. In addition, the total length of stay in days and overall cost of stay would also be estimated and compared between the two study arms. These secondary objectives are purely descriptive and no hypothesis testing is planned for these objectives.

Randomization schedule will be generated using standard statistical software by a statistician who is not going to be involved in data analysis. Envelopes containing the treatment instructions will be marked according to that schedule. Randomization will be performed in blocks of six subjects, three for intervention and three for control arm, to ensure balanced groups.

If the proposed algorithm is validated and found to be of value, it can potentially be implemented nationwide as a standard protocol for the evaluation of suspected appendicitis. This may reduce the number of unwarranted CT scans performed and reduce health care costs. In addition, the reduction of unnecessary CT scans helps to minimize unwarranted radiation exposure which is not insignificant. A single CT Abdomen Pelvis for evaluation of suspected appendicitis exposes one to 14 mSv of ionizing radiation which adds an additional cancer risk of up to 0.2% for an individual who is 30 years of age. The cumulative effects of such radiation exposure may prove significant and a management algorithm guiding sensible CT utilization will help ease the burden of radiation induced complications in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 21 to 80 who are admitted to Singapore General Hospital and Sengkang Health for suspected appendicitis based on admission diagnosis from the Emergency Department

Exclusion Criteria:

* Patients who are pregnant
* Patients below 21 or above 80 years of age
* Patients with generalized peritonitis on presentation
* Patients with palpable right iliac fossa mass on presentation
* Patients with evidence of acute confusional state/dementia
* Patients at high risk of surgery (ASA>4) from the study
* Patients who are immunocompromised (on chemotherapy, steroids etc.)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of CT performed | Through study completion, an average of 2 years.
  The percentage of CT scans performed for patients within each management arm

SECONDARY OUTCOMES:
Percentage of negative appendectomy | Through study completion, an average of 2 years.
  Patients who were operated with a pre-operative diagnosis of acute appendicitis with subsequent histology showing no features of acute appendicitis
Percentage of missed diagnosis | 2 weeks after discharge
  Patients who were not diagnosed with acute appendicitis during the initial admission but were subsequently readmitted within 2 weeks of discharge due to progression of symptoms, with eventual surgery showing acute appendicitis on histology.
Length of stay | 2 weeks after discharge
  Duration of total hospitalization (measured in days) from point of admission to discharge.
Cost of stay | 2 weeks after discharge
  Total cost of stay incurred by the patient in Singapore Dollars during admission before government subsidies were taken into consideration

CONTACTS AND LOCATIONS:
Overall Officials: Tan Jianhong Winson, MBBS, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - Sengkang Health, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birnbaum BA, Wilson SR. Appendicitis at the millennium. Radiology. 2000 May;215(2):337-48. doi: 10.1148/radiology.215.2.r00ma24337. PMID 10796905
- [Background] Rothrock SG, Pagane J. Acute appendicitis in children: emergency department diagnosis and management. Ann Emerg Med. 2000 Jul;36(1):39-51. doi: 10.1067/mem.2000.105658. PMID 10874234
- [Background] Yildirim E, Karagulle E, Kirbas I, Turk E, Hasdogan B, Teksam M, Coskun M. Alvarado scores and pain onset in relation to multislice CT findings in acute appendicitis. Diagn Interv Radiol. 2008 Mar;14(1):14-8. PMID 18306139
- [Background] Hong JJ, Cohn SM, Ekeh AP, Newman M, Salama M, Leblang SD; Miami Appendicitis Group. A prospective randomized study of clinical assessment versus computed tomography for the diagnosis of acute appendicitis. Surg Infect (Larchmt). 2003 Fall;4(3):231-9. doi: 10.1089/109629603322419562. PMID 14588157
- [Background] Jones K, Pena AA, Dunn EL, Nadalo L, Mangram AJ. Are negative appendectomies still acceptable? Am J Surg. 2004 Dec;188(6):748-54. doi: 10.1016/j.amjsurg.2004.08.044. PMID 15619494
- [Background] Smink DS, Finkelstein JA, Garcia Pena BM, Shannon MW, Taylor GA, Fishman SJ. Diagnosis of acute appendicitis in children using a clinical practice guideline. J Pediatr Surg. 2004 Mar;39(3):458-63; discussion 458-63. doi: 10.1016/j.jpedsurg.2003.11.015. PMID 15017570
- [Background] Berrington de Gonzalez A, Darby S. Risk of cancer from diagnostic X-rays: estimates for the UK and 14 other countries. Lancet. 2004 Jan 31;363(9406):345-51. doi: 10.1016/S0140-6736(04)15433-0. PMID 15070562
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Brenner DJ. Minimising medically unwarranted computed tomography scans. Ann ICRP. 2012 Oct-Dec;41(3-4):161-9. doi: 10.1016/j.icrp.2012.06.004. Epub 2012 Aug 22. PMID 23089015
- [Background] Alvarado A. A practical score for the early diagnosis of acute appendicitis. Ann Emerg Med. 1986 May;15(5):557-64. doi: 10.1016/s0196-0644(86)80993-3. PMID 3963537
- [Background] National Research Council (US) Board on Radiation Effects Research. Health Risks from Exposure to Low Levels of Ionizing Radiation: BEIR VII, Phase I, Letter Report (1998). Washington (DC): National Academies Press (US); 1998. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK224187/ PMID 25077203
- [Background] Mettler FA Jr, Huda W, Yoshizumi TT, Mahesh M. Effective doses in radiology and diagnostic nuclear medicine: a catalog. Radiology. 2008 Jul;248(1):254-63. doi: 10.1148/radiol.2481071451. PMID 18566177
- [Derived] Tan WJ, Acharyya S, Chew MH, Foo FJ, Chan WH, Wong WK, Ooi LL, Ng JCF, Ong HS. Randomized control trial comparing an Alvarado Score-based management algorithm and current best practice in the evaluation of suspected appendicitis. World J Emerg Surg. 2020 May 1;15(1):30. doi: 10.1186/s13017-020-00309-0. PMID 32357897